CLINICAL TRIAL: NCT01399580
Title: A Phase 2b, Prospective, Double-Blind, Placebo-Controlled, Multicenter Study to Evaluate Efficacy and Safety of Atrasentan, Including Thoracic Bioimpedance, in Type 2 Diabetic Subjects With Nephropathy
Brief Title: A Prospective, Double-Blind, Placebo-Controlled, Multicenter Study to Evaluate Efficacy and Safety of Atrasentan, Including Thoracic Bioimpedance, in Type 2 Diabetic Subjects With Nephropathy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AbbVie (prior sponsor, Abbott) (Industry)
Responsible Party: Sponsor
Organization: AbbVie (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: M12-830
Record Dates: First submitted 2011-07-20; First posted 2011-07-22 (Estimated); Last update posted 2013-10-25 (Estimated); Status verified 2013-09

CONDITIONS: Chronic Kidney Disease; Diabetic Nephropathy
Keywords: endothelin receptor antagonists
MeSH Terms: conditions — Renal Insufficiency, Chronic; Diabetic Nephropathies | interventions — Atrasentan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Group A - Placebo QD (Placebo Comparator)
  Interventions: Drug: Placebo
- Group B - Low dose Atrasentan QD (Active Comparator)
  Interventions: Drug: Atrasentan
- Group C - High dose Atrasentan QD (Active Comparator)
  Interventions: Drug: Atrasentan

INTERVENTIONS:
Drug: Atrasentan — Subjects will take two tablets daily of either low dose Atrasentan QD or high dose Atrasentan QD for 8 weeks during the treatment period.
  Other Names: ABT-627
  Arms: Group B - Low dose Atrasentan QD; Group C - High dose Atrasentan QD
Drug: Placebo — Subjects will take two tablets daily of placebo QD for 8 weeks during the treatment period.
  Arms: Group A - Placebo QD

SUMMARY:
Prospective, Randomized, Double-Blind, Parallel Design, Placebo-Controlled Multicenter Study. The study objectives are to evaluate efficacy and safety, including thoracic bioimpedance, of once daily administration of atrasentan tablets (high dose and low dose) compared to placebo in type 2 diabetic subjects with nephropathy who are receiving the maximum tolerated labeled daily dose of a RAS inhibitor.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is greater than or equal to 18 years old.
2. Subject has type 2 diabetes and has been treated with at least one anti-hyperglycemic medication within the 12 months prior to the Screening Period.
3. Subject is currently receiving an angiotensin converting enzyme inhibitor (ACEi) or Angiotensin II receptor blocker (ARB) (Renin Angiotensin System (RAS) inhibitor).
4. If female, subject is not breastfeeding and is not pregnant (verified by negative serum pregnancy test prior to the Treatment Period). Subject is not of childbearing potential, defined as postmenopausal for at least one year or surgically sterile (bilateral tubal ligation, bilateral oophorectomy or hysterectomy) or is of childbearing potential and practicing one of the approved methods of birth control as defined in the Clinical Trial Protocol. Contraception must be used during the study and for 4 weeks after the last dose of study drug.
5. For entry into the Run-in Period the subject must satisfy the following criteria based on the Screening laboratory values:

   * Estimated glomerular filtration rate (eGFR) greater than or equal to 30 and less than or equal to 75 mL/min/1.73m^2 by the Epidemiology Collaboration (EPI) formula
   * Urinary Albumin to Creatinine Ratio (UACR) greater than or equal to 300 and less than or equal to 3500 mg/g as determined by the geometric mean of the two morning void urine specimens obtained at the Screening visit
   * Serum albumin greater than or equal to 3.0 g/dL
   * B-Type Natriuretic Peptide (BNP) less than or equal to 200 pg/mL
   * Negative serum pregnancy test for female subjects
   * Systolic Blood Pressure (SBP) greater than or equal to 110 mmHg and less than or equal to 180 mmHg
   * Glucosylated hemoglobin (HbA1c) less than or equal to 12%
6. For entry into the Treatment Period the subject must satisfy the following criteria based on the last visit of the Run-in Period laboratory values:

   * Renin Angiotensin System (RAS) inhibitor at maximum tolerated labeled dose for the previous 4 weeks with no adjustment of dose
   * Diuretic at any dose unless medically contraindicated (with the exception of loop diuretics greater than or equal to 120 mg QD of furosemide or greater than or equal to 3.0 mg QD of bumetanide or greater than or equal to 150 mg QD of ethacrynic acid or greater than or equal to 60 mg QD of torasemide)
   * UACR ≥ 200 mg/g as determined by the median of the three morning void urine specimens obtained prior to the Week -1 visit
   * Systolic Blood Pressure (SBP) greater than or equal to 110 mmHg and less than or equal to 160 mmHg
   * Serum Potassium less than or equal to 5.5 mEq/L
   * Negative serum pregnancy test for female subjects

Exclusion Criteria:

1. Patient has a history of moderate or severe edema, facial edema unrelated to trauma, or a history of myxedema in the prior 6 months to Screening.
2. Subject is receiving loop diuretics greater than or equal to 120 mg QD of furosemide or greater than or equal to 3.0 mg QD of bumetanide or greater than or equal to 150 mg QD of ethacrynic acid or greater than or equal to 60 mg QD of torasemide.
3. Subject has a history of pulmonary edema.
4. Subject has a history of pulmonary hypertension, or any lung diseases requiring oxygen therapy (i.e., chronic obstructive pulmonary disease, emphysema, pulmonary fibrosis).
5. Subject has a history of orthostatic hypotension within the past 6 months as defined by the presence of a supine-to-standing blood pressure decrease greater than or equal to 20 mmHg systolic or greater than or equal to 10 mmHg diastolic within 3 minutes of standing.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2011-08; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Change from baseline to each post-baseline visit up to Week 8 in log-transformed Urinary Albumin to Creatinine Ratio (UACR) | Every two weeks for 8 weeks

SECONDARY OUTCOMES:
Change from baseline to each post baseline measure for estimated glomerular filtration rate (eGFR) | Every two weeks for 8 weeks
The change from baseline to each post-baseline assessment of thoracic bioimpedance | Treatment Day 1, Week 1, 2, 4, 6, 8 and 30 days post-treatment

CONTACTS AND LOCATIONS:
Overall Officials: Blai Coll, MD, Study Director — AbbVie
Locations (28):
- United States (28):
  - Site Reference ID/Investigator# 58144, Phoenix, Arizona
  - Site Reference ID/Investigator# 71034, Tempe, Arizona
  - Site Reference ID/Investigator# 56927, Azusa, California
  - Site Reference ID/Investigator# 70793, Azusa, California
  - Site Reference ID/Investigator# 64027, Chula Vista, California
  - Site Reference ID/Investigator# 54120, Concord, California
  - Site Reference ID/Investigator# 64026, La Mesa, California
  - Site Reference ID/Investigator# 70173, Los Angeles, California
  - Site Reference ID/Investigator# 54121, Denver, Colorado
  - Site Reference ID/Investigator# 56924, Boynton Beach, Florida
  - Site Reference ID/Investigator# 56642, Hollywood, Florida
  - Site Reference ID/Investigator# 68986, Augusta, Georgia
  - Site Reference ID/Investigator# 56644, Chicago, Illinois
  - Site Reference ID/Investigator# 54129, Baton Rouge, Louisiana
  - Site Reference ID/Investigator# 68982, Pontiac, Michigan
  - Site Reference ID/Investigator# 64023, Albany, New York
  - Site Reference ID/Investigator# 55543, Flushing, New York
  - Site Reference ID/Investigator# 54164, Fargo, North Dakota
  - Site Reference ID/Investigator# 58147, Willoughby Hills, Ohio
  - Site Reference ID/Investigator# 54123, Bethlehem, Pennsylvania
  - Site Reference ID/Investigator# 61742, Pittsburgh, Pennsylvania
  - Site Reference ID/Investigator# 54132, Chattanooga, Tennessee
  - Site Reference ID/Investigator# 54108, Dallas, Texas
  - Site Reference ID/Investigator# 54126, Greenville, Texas
  - Site Reference ID/Investigator# 58153, Houston, Texas
  - Site Reference ID/Investigator# 54110, Houston, Texas
  - Site Reference ID/Investigator# 54116, North Richland Hills, Texas
  - Site Reference ID/Investigator# 54173, Silverdale, Washington

REFERENCES:
- [Derived] Lin CW, Mostafa NM, L Andress D, J Brennan J, Klein CE, Awni WM. Relationship Between Atrasentan Concentrations and Urinary Albumin to Creatinine Ratio in Western and Japanese Patients With Diabetic Nephropathy. Clin Ther. 2018 Feb;40(2):242-251. doi: 10.1016/j.clinthera.2017.07.011. Epub 2017 Jul 27. PMID 28756065